CLINICAL TRIAL: NCT04279119
Title: An Open Label, Phase 1, Maximal Usage Pharmacokinetics and Safety Study of ARQ-151 Cream 0.3% Administered QD in Adolescent and Adult Subjects With Chronic Plaque Psoriasis
Brief Title: Maximal Usage Pharmacokinetics and Safety of ARQ-151 in Adolescents and Adults With Chronic Plaque Psoriasis
Acronym: MUSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-107
Record Dates: First submitted 2020-01-15; First posted 2020-02-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 cream 0.3% (Experimental): Open label study of ARQ-151 cream 0.3% applied once daily for 2 weeks
  Interventions: Drug: ARQ-151- cream 0.3%

INTERVENTIONS:
Drug: ARQ-151- cream 0.3% — ARQ-151 cream 0.3% applied to chronic plaque psoriasis lesions once a day for 2 weeks

SUMMARY:
This is a phase 1, open label, single arm study in which ARQ-151 cream 0.3% is applied QD for 2 weeks to adolescent subjects with chronic plaque psoriasis involving at least 10% body surface area (BSA) and adult subjects with chronic plaque psoriasis involving at least 20% BSA (excluding scalp).

The objectives of this study are to evaluate the exposure and characterize the plasma pharmacokinetic profile and to assess the safety and tolerability of ARQ-151 cream 0.3% administered once daily for 2 weeks to adolescent and adult subjects with chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent or for adolescents assent with consent of a parent or legal guardian.
2. Males and females ages 12 years and older (inclusive) at the time of consent/assent.
3. Clinical diagnosis of psoriasis vulgaris of at least 3 months duration as determined by the Investigator or through subject interview. Stable disease for the past 4 weeks.
4. Psoriasis vulgaris on the face, extremities, trunk, and/or intertriginous areas involving at least 10% of BSA in adolescents and at least 20% of BSA in adults (excluding the scalp).
5. An Investigator Global Assessment of disease severity of at least Moderate ('3') at Baseline.
6. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial.
7. Females of non-childbearing potential should be premenarchal, post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.
8. Subjects in good health as judged by the Investigator, based on medical history, physical examination, vital signs, 12-lead electrocardiogram, serum chemistry labs, hematology values, and urinalysis.
9. Subjects are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects who cannot discontinue medication and treatments prior to the Baseline visit and during the study according to Excluded Medications and Treatments (Table 1).
2. Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other light emitting diode (LED).
3. Subjects currently taking lithium or antimalarial drugs.
4. Planned initiation or changes to concomitant medication that could, in the opinion of the Investigator, affect psoriasis vulgaris (e.g. beta blockers, ACE inhibitors).
5. Current diagnosis of non-plaque form of psoriasis (e.g., guttate, erythrodermic/exfoliative, or pustular psoriasis). Current diagnosis of drug-induced psoriasis.
6. Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
7. Known allergies to excipients in ARQ-151 cream
8. Subjects who cannot discontinue the use of systemic strong P 450 cytochrome inhibitors (e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, fluconazole, nefazodone, saquinavir, suboxone and telithromycin) for two weeks prior to the Baseline visit and during the study period.
9. Subjects who cannot discontinue the use of systemic strong P 450 cytochrome inducers (e.g., efavirenz, nevirapine, glucocorticoids, barbiturates (including phenobarbital), phenytoin, rifampin and carbamazepine) for two weeks prior to the Baseline visit and during the study period.
10. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
11. Subjects who have received oral roflumilast (Daliresp®, Daxas®) or other PDE4 inhibitors (apremilast) within the past 4 weeks.
12. Known or suspected:

    * severe renal insufficiency or moderate to severe liver impairment (Child-Pugh B or C)
    * known HIV infection
    * hypersensitivity to component(s) of the investigational products
    * history of severe depression, suicidal ideation, Baseline/Screening C-SSRS indicative of suicidal ideation, whether lifetime or recent/current
13. Adult subjects with PHQ-8 ≥10 or adolescent subjects with modified PHQ-A ≥10 at Screening or Baseline visits.
14. Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of investigational product.
15. Subjects with a history of a major surgery within 4 weeks prior to Baseline (Visit 2) or has a major surgery planned during the study.
16. Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation. For adolescent subjects; parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language.
17. Subjects who are family members of the clinical study site, clinical study staff, or Sponsor.
18. Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
19. Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
20. Subjects with active infection that required oral or intravenous administration of antibiotics, antifungal or antiviral agents within 7 days of Baseline/Day 1.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of roflumilast and its major N-oxide metabolite | 5 weeks
  Maximum observed concentration of drug in plasma metabolite
Area under the plasma concentration-time curve until the last quantifiable timepoint (AUC) for roflumilast and its N-oxide metabolite | 5 weeks
  The area under the plasma concentration-time curve (AUC) is a method of measurement of the total exposure of a drug in plasma.
Time of maximum concentration (Tmax) of roflumilast and its major N-oxide metabolite | 5 weeks
  Tmax is the time that a drug achieves maximum concentration in plasma

SECONDARY OUTCOMES:
Subject incidence of adverse events | 5 weeks
  Number of participants with adverse events during treatment will be assessed
Incidence of application site reactions | 5 weeks
  Number of subjects that experience an application site skin reaction by investigator assessment and application site reactions reported as adverse events will be assessed
Incidence of application site reactions | 5 weeks
  Percentage of subjects that experience an application site skin reaction by investigator assessment and application site reactions reported as adverse events will be assessed
The incidence of suicide ideation as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | 5 weeks
  The C-SSRS is a tool used to assess suicide risk, the severity and immediacy of that risk. The C-SSRS is made up of ten categories and includes questions that require binary responses (yes/no) to indicate a presence or absence of the behavior and follow-up questions for any behavior that is endorsed (yes) to collect additional information.
The incidence of changes from baseline in the Patient Health Questionnaire (PHQ-8) Depression Scale | 5 weeks
  The PHQ-8 is an instrument used for screening, diagnosing, monitoring and measuring the severity of depression in adults. The score for the PHQ-8 ranges from 0-24 with a higher score reflecting a higher severity category of depression.
The incidence of changes from baseline in the Patient Health Questionnaire for Adolescents (PHQ-A) Depression Scale | 5 weeks
  The PHQ-A is an instrument used for screening, diagnosing, monitoring and measuring the severity of depression in adolescents. The score for the PHQ-A ranges from 0-24 with a higher score reflecting a higher severity category of depression.

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (12):
- United States (12):
  - Arcutis Clinical Site 09, Rogers, Arkansas
  - Arcutis Clinical Site 11, Fountain Valley, California
  - Arcutis Clinical Site 07, Coral Gables, Florida
  - Arcutis Clinical Site 03, Doral, Florida
  - Arcutis Clinical Site 06, Hialeah, Florida
  - Arcutis Clinical Site 12, Miami, Florida
  - Arcutis Clinical Site 04, Sanford, Florida
  - Arcutis Clinical Site 02, Plainfield, Indiana
  - Arcutis Clinical Site 01, Dublin, Ohio
  - Arcutis Clinical Site 10, Arlington, Texas
  - Arcutis Clinical Site 05, San Antonio, Texas
  - Arcutis Clinical Site 08, Richmond, Virginia

REFERENCES:
- [Derived] Thurston AW Jr, Osborne DW, Snyder S, Higham RC, Burnett P, Berk DR. Pharmacokinetics of Roflumilast Cream in Chronic Plaque Psoriasis: Data from Phase I to Phase III Studies. Am J Clin Dermatol. 2023 Mar;24(2):315-324. doi: 10.1007/s40257-022-00741-9. Epub 2022 Nov 24. PMID 36422852